CLINICAL TRIAL: NCT06993844
Title: A Phase 1/2, Open-label, First-in-human Study of the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ETX-636, a Pan-mutant-selective PI3Kα Inhibitor, as Monotherapy and in Combination With Other Anticancer Therapies in Participants With Advanced Solid Tumors
Brief Title: Phase 1/2 Study of ETX-636 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ensem Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ETX636-C-001
Record Dates: First submitted 2025-05-01; First posted 2025-05-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors; Advanced Breast Cancer
Keywords: cancer; breast cancer; solid tumors; PIK3CA; PI3Kα inhibitor; Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; HER2-negative breast cancer; HR-positive breast cancer; Gynecologic cancer; Endometrial cancer; Ovarian cancer; Cervical cancer; Head and neck cancer; Head and neck squamous cell carcinoma; Fulvestrant; Antineoplastic Agents; PI3Kα; PI3K alpha; PI3Kα mutation; Alpelisib; Estrogen Receptor Antagonists; Estrogen Antagonists; Hormone Receptor Antagonists; Hormone Antagonists; Hormones, Hormone Substitutes, and Hormone Antagonists; Physiological Effects of Drugs; PIK3CA mutation
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Hereditary Sensory and Autonomic Neuropathies; Neoplasms by Site; Breast Diseases; Endometrial Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Fulvestrant

STUDY DESIGN:
Intervention Model Description: Fulvestrant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A Dose Escalation Monotherapy (Advanced Solid Tumors with PIK3CA mutation) (Experimental): Part A is a dose escalation monotherapy of ETX-636 in advanced solid tumors with PIK3CA mutation
  Interventions: Drug: ETX-636 dose escalation
- Part B Dose Escalation Combination Therapy (HR+/HER2- locally advanced or metastatic breast cancer) (Experimental): Part B is a dose escalation combination therapy in HR+/HER2- locally advanced or metastatic breast cancer. The study treatment will be ETX-636, a pan-mutant-selective PI3Kα inhibitor, in combination with fulvestrant (Faslodex) at a fixed dose of 500 mg IM.
  Interventions: Drug: ETX-636 dose escalation in combination with fulvestrant
- Part C Dose Expansion Combination Therapy (HR+/HER2- locally advanced or metastatic breast cancer) (Experimental): Part B is a dose expansion combination therapy in HR+/HER2- locally advanced or metastatic breast cancer. The study treatment will be ETX-636, a pan-mutant-selective PI3Kα inhibitor, in combination with fulvestrant (Faslodex) at a fixed dose of 500 mg IM.
  Interventions: Drug: ETX-636 dose expansion in combination with fulvestrant

INTERVENTIONS:
Drug: ETX-636 dose escalation — ETX-636 is a pan-mutant-selective PI3Kα Inhibitor and degrader in the form of an oral tablet that will be taken once per day in 28-day cycles, to evaluate escalating dose levels.
  Arms: Part A Dose Escalation Monotherapy (Advanced Solid Tumors with PIK3CA mutation)
Drug: ETX-636 dose escalation in combination with fulvestrant — ETX-636 is a pan-mutant-selective PI3Kα Inhibitor and degrader in the form of an oral tablet. ETX-636 will be taken in combination with fulvestrant in 28-day cycles, to evaluate escalating dose levels. EXT-636 is an oral tablet that will be taken once per day. Fulvestrant will be administered as an injection 2 weeks apart in the first 28 days, followed by monthly injections.
  Other Names: Faslodex
  Arms: Part B Dose Escalation Combination Therapy (HR+/HER2- locally advanced or metastatic breast cancer)
Drug: ETX-636 dose expansion in combination with fulvestrant — ETX-636 is a pan-mutant-selective PI3Kα Inhibitor and degrader in the form of an oral tablet. ETX-636 will be taken in combination with fulvestrant in 28-day cycles, to expand selected dose levels. EXT-636 is an oral tablet that will be taken once per day. Fulvestrant will be administered as an injection 2 weeks apart in the first 28 days, followed by monthly injections.
  Other Names: Faslodex
  Arms: Part C Dose Expansion Combination Therapy (HR+/HER2- locally advanced or metastatic breast cancer)

SUMMARY:
Phase 1/2, open-label study of ETX-636 in participants with advanced solid tumors

DETAILED DESCRIPTION:
Brief Summary: This is a Phase 1/2, open-label, multicenter, 3-part study to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of ETX-636 in participants with advanced solid tumors harboring a PIK3CA mutation.

Part A will evaluate escalating doses of ETX-636 as monotherapy in participants with advanced solid tumors. Part B will evaluate escalating doses of ETX-636 as combination therapy with fixed dose fulvestrant in participants with hormone receptor positive (HR+), HER2 negative (HER2-) locally advanced or metastatic breast cancer. Part C will be a combination therapy expansion in participants with HR+, HER2- locally advanced or metastatic breast cancer.

Each study part will include a 28-day screening period, followed by treatment with ETX-636 monotherapy or combination therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Metastatic or locally advanced and unresectable solid tumor that has progressed on or after at least one available therapy.
* Tumor harboring an activating PIK3CA mutation detected in either tumor tissue or ctDNA.
* At least 1 measurable lesion or evaluable disease per RECIST v1.1.
* An ECOG performance status score of 0 or 1.
* Adequate organ function.

Additional key inclusion criterion for Parts B and C:

- Confirmed metastatic or locally advanced HR+/HER2- breast cancer not amenable to surgical resection with curative intent and must have received at least 1 prior CDK4/6 inhibitor and at least 1 prior anti-estrogen therapy.

Key Exclusion Criteria:

* Has history (within ≤2 years before screening) of a solid tumor or hematological malignancy that is histologically distinct from the cancers being studied.
* Has symptomatic brain or spinal metastases or a known or suspected history of untreated or uncontrolled central nervous system (CNS) involvement.
* Has an established diagnosis of diabetes mellitus type 1 or has uncontrolled diabetes mellitus type 2.
* Has received treatment with any local or systemic anticancer therapy or investigational anticancer agent within 14 days prior to start of treatment.
* Has toxicities from previous anticancer therapies that have not resolved to baseline levels with the exception of alopecia and peripheral neuropathy.
* Has had radiotherapy outside the target tumor lesions within 14 days prior to start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate Safety and Tolerability of ETX-636 monotherapy in Part A and ETX-636 plus fulvestrant combination therapy in Part B | First 28 days of treatment
  Proportion of participants who experience at least 1 Dose Limiting Toxicity (DLT)
Evaluate Safety and Tolerability of ETX-636 monotherapy in Part A and ETX-636 plus fulvestrant combination therapy in Part B | Average of 6 months
  Incidence of AEs, treatment discontinuations due to AEs, changes from baseline in laboratory assessments, ECGs and vital signs.
Select the Recommended Phase 2 Dose(s) (RP2D) in Part B to be further explored in Part C (combination therapy expansion) | Average of 6 months
  Safety Parameters as described for primary outcomes
Evaluate efficacy of ETX-636 plus fulvestrant combination therapy at the RP2D(s) in Part C | Average of 6 months
  ORR and CBR according to RECIST v1.1

SECONDARY OUTCOMES:
Characterize the Cmax (PK) of ETX-636 monotherapy in Part A and ETX-636 plus fulvestrant combination therapy in Part B | First 2 treatment cycles (each cycle is 28 days)
  Maximum observed plasma concentration (Cmax) of ETX-636
Characterize the Tmax (PK) of ETX-636 monotherapy in Part A and ETX-636 plus fulvestrant combination therapy in Part B | First 2 treatment cycles (each cycle is 28 days)
  Calculated time to reach maximum observed plasma concentration of ETX-636
Characterize the AUC (PK) of ETX-636 monotherapy in Part A and ETX-636 plus fulvestrant combination therapy in Part B | First 2 treatment cycles (each cycle is 28 days)
  Calculated area under the plasma concentration curve (AUC) of ETX-636
Measure PD effects of ETX-636 monotherapy in Part A and ETX-636 plus fulvestrant combination therapy in Part B and ETX-636 plus fulvestrant at the RP2D(s) in Part C | First 3 cycles (each cycle is 28 days)
  Change from baseline in ctDNA levels; Change from baseline in PD markers in paired biopsies
Changes in fasting blood glucose (All Parts) | Average of 6 months
  Measured by fasting blood glucose
Changes in longitudinal glucose metabolism (All Parts) | Average of 6 months
  Measured by HbA1c
Assess preliminary efficacy of ETX-636 monotherapy in Part A and ETX-636 plus fulvestrant combination therapy in Part B | Average of 6 months
  Objective response rate (ORR) and clinical benefit rate (CBR) based on RECIST v1.1
Evaluate measures of efficacy of ETX-636 plus fulvestrant combination therapy at the RP2D(s) in Part C | Average of 6 months
  Time to response (TTR) according to RECIST v1.1
Evaluate additional measures of efficacy of ETX-636 plus fulvestrant combination therapy at the RP2D(s) in Part C | Average of 6 months
  Duration of response (DoR) according to RECIST v1.1
Evaluate additional measures of efficacy of ETX-636 plus fulvestrant combination therapy at the RP2D(s) in Part C | Average of 6 months
  Disease control rate (DCR) according to RECIST v1.1
Evaluate additional measures of efficacy of ETX-636 plus fulvestrant combination therapy at the RP2D(s) in Part C | Average of 6 months
  Progression free survival (PFS) according to RECIST v1.1
Evaluate Safety of ETX-636 plus fulvestrant combination therapy at the RP2Ds in Part C | Average of 6 months
  Incidence of adverse events graded according to CTCAE v5.0
Evaluate tolerability of ETX-636 plus fulvestrant combination therapy at the RP2Ds in Part C | Average of 6 months
  Incidence of adverse events graded according to CTCAE v5.0
Characterize the PK of ETX-636 plus fulvestrant using population PK modeling (Part C, to be reported separately) | First 2 treatment cycles (each cycle is 28 days)
  Plasma concentrations

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - START, San Antonio, Texas
  - NEXT, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided